CLINICAL TRIAL: NCT03030430
Title: Randomized, Double-blind, Single-dose, 3-arm Parallel Design Comparative Pharmacokinetic(PK) and Safety Study of BAT1706 Versus European Union(EU)-Sourced Avastin® and United State (US)-Sourced Avastin® Administered in Healthy Subjects
Brief Title: Study of Bevacizumab(BAT1706) and Comparators in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-1706-001
Record Dates: First submitted 2017-01-20; First posted 2017-01-25 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: NSCLC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- BAT1706 (Experimental): BAT1706 injection
  Interventions: Biological: BAT1706 injection
- EU-sourced Avastin (Active Comparator): EU-sourced Avastin
  Interventions: Biological: EU-sourced Avastin
- US-sourced Avastin (Active Comparator): US-sourced Avastin
  Interventions: Biological: US-sourced Avastin

INTERVENTIONS:
Biological: BAT1706 injection — 1mg/kg, IV on day 1
  Arms: BAT1706
Biological: EU-sourced Avastin — 1mg/kg, IV on day 1
  Arms: EU-sourced Avastin
Biological: US-sourced Avastin — 1mg/kg, IV on day 1
  Arms: US-sourced Avastin

SUMMARY:
The purpose of this study is to establish PK similarity in the treatment of BAT1706 and comparators.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, single-dose, 3-arm parallel group study to compare the PK, and to evaluate the safety, tolerability and immunogenicity, of BAT1706, EU-Avastin and US-Avastin after a single IV infusion in healthy adult male subjects.

A total of 129 healthy male subjects who meet the required entry criteria will be randomly assigned to one of three treatment groups in a 1:1:1 ratio to receive a single IV infusion of either BAT1706, EU-Avastin or US-Avastin. A total of 117 evaluable subjects are required.

Initially, subjects will be administered the study drug in staggered groups; the first group will comprise 3 subjects, the second group 6 subjects and the third group 9 subjects. Within each group subjects will be randomized to ensure equal numbers of subjects receive each of the three treatments.

There will be at least 48 hours between administrations of study drug to each group. Prior to administration of study drug to the next group, the safety and tolerability findings of the preceding group will be reviewed by the Principal Investigator. The next group will be dosed provided there are no serious or unexpected drug-related safety issues. Each subject will be required to remain in the clinical center for 48 hours after dosing for safety evaluation.

After the first 3 groups have been evaluated, the Principal Investigator will decide whether to proceed with continuous enrolment according to the clinical center capability.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males aged 18 to 50 years inclusive and body weight 65 to 100kg.
2. Subjects who are healthy as determined by pre-study medical history, physical examination, vital signs and 12 ECG.
3. Subjects whose clinical laboratory test results are normal, or where outside the reference range are judged as not clinical relevant.

Exclusion Criteria:

1. Have a history of and/or current clinically significant gastrointestinal, renal, hepatic, cardiovascular, haematological, pulmonary, neurologic, metabolic, psychiatric or allergic disease excluding mild asymptomatic seasonal allergies.
2. Subject with a psychiatric disorder or considered unsuitable for inclusion by the investigator.
3. History or current clinically significant, excluding mild asymptomatic seasonal allergies, hypersensitivity or allergic reactions including known or suspected drug hypersensitivity to any component of the study drug formulations or comparable drugs.
4. Any biological drug within 3 months or monoclonal antibodies within 9 months of study drug administration.
5. Intake of herbal remedies within 14 days prior to study drug administration.
6. History of alcohol abuse or a positive alcohol test on screening or admission to the clinical center.
7. Any persons who are:an employee of the Principal Investigator, clinical center, Clinical Research Organization (CRO) or Sponsor;a relative of an employee of the clinical center, the Investigators, CRO or the Sponsor.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
area under curve (AUC)0~∞ | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Chris Wynne, Medical Doc, Principal Investigator — Director
Locations (1):
- Christchurch Clinical Studies Trust Ltd (CCST), Christchurch, New Zealand

REFERENCES:
- [Derived] Wu X, Wynne C, Xu C, Gan Y, Wang C, Thomas BE, Yu JC, Li S, Zhang L. A Global Phase I Clinical Study Comparing the Safety and Pharmacokinetics of Proposed Biosimilar BAT1706 and Bevacizumab (Avastin(R)) in Healthy Male Subjects. BioDrugs. 2019 Jun;33(3):335-342. doi: 10.1007/s40259-019-00352-7. PMID 31016568